CLINICAL TRIAL: NCT06670456
Title: Multicentral Observational Prospective Cohort of Patients With Spontaneous Intracerebral Hemorrhage
Brief Title: Prospective Cohort of Patients With Intracerebral Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: De-zhi Kang (Other)
Collaborators: Fuzhou University (Other); Fujian Medical University (Other); National Institute of Hospital Administration (China) (Unknown)
Responsible Party: Sponsor-Investigator, De-zhi Kang, Prof., First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: 2022ZD01003
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Acute; Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — 1. Peripheral blood; 2. Cerebrospinal fluid; 3. Evacuated hematoma, cerebral tissue, and/or bone flap. (No for everyone)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators designed a multicentral, observational, prospective cohort study to provide cortical data for risk stratification and biomarkers on early outcomes, complications, long-term neurological function, and cognitive status of spontaneous intracerebral hemorrhage patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spontaneous intracerebral hemorrhage (ICH) through skull radiologic scans (CT or MRI);
* Underwent no surgical intervention;

Exclusion Criteria:

* Secondary intracerebral hemorrhage (with leading cause, e.g., Moyamoya disease, arteriovenous malformation, intracranial aneurysm, tumor, brain trauma)
* Pre-stroke life expectancy < 1 year for severe comorbidities (e.g., Progressive malignant tumor, severe chronic heart failure [NYHA: III-IV], severe chronic obstructive pulmonary disease [III-IV], chronic kidney disease requiring hemodialysis)
* Severe dependency or incorporation to interview (e.g., pre-stroke mRS>3, severe dementia, intractable mental disease)
* Unsuitable for inclusion in the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with spontaneous intracerebral hemorrhage and received no surgical intervention until enrollment; and those patients should have enough life expectancy and be assessable for the interview, according to their pre-stroke status.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Neurological Function | Discharge; 3, 6, 12 months after enrollment
  Assessed with modified Rankin Scale (0-6)
Mortality | Discharge; 3, 6, 12 months after enrollment

SECONDARY OUTCOMES:
Complications | Admission period; the 3, 6, 12 months after enrollment
  Lately stoke, epilepsy, infections, cardiac event, ebolism.
Cognitive Status | The 3, 6, 12 months after enrollment
  Assessed with Telephone Interview for Cognitive Status - Modifed scale (0-51) Chinese version

CONTACTS AND LOCATIONS:
Overall Officials: De-zhi Kang, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (6):
- China (6):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Anxi County Hospital, Quanzhou, Fujian
  - Jinjiang Municipal Hospital, Quanzhou, Fujian
  - The Second Affiliated lospital of Xiamen Medical College, Xiamen, Fujian
  - Zhangzhou Municipal Hospital, Zhangzhou, Fujian
  - Liaocheng People's Hospital, Liaocheng, Shandong

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified case data are available from the authors upon reasonable request, after request in writing to the corresponding authors and after approval by the study committee and principal investigators from each site.